CLINICAL TRIAL: NCT02406677
Title: Affordability and Real-world Antiplatelet Treatment Effectiveness After Myocardial Infarction Study
Acronym: ARTEMIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: D5130R00030
Record Dates: First submitted 2015-03-30; First posted 2015-04-02 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Cost Sharing, Acute Coronary Syndrome
Keywords: Acute Coronary Syndromes, ACS, Myocardial Infarction, STEMI, NSTEMI, MI, Co-Payments, Copay, Cost Sharing
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Copayment Intervention Arm (Experimental): Sites in the intervention arm will provide patients with a study voucher card to offset any patient copayments or medication card for the filling of any prescriptions of clopidogrel or ticagrelor.
  Interventions: Other: Study voucher card
- Usual Care Arm (No Intervention): For hospitals randomized to the control arm, all patients receive usual care and no study intervention is performed.

INTERVENTIONS:
Other: Study voucher card — Study voucher card to offset any patient copayments or medication costs for the filling of any prescriptions of clopidogrel or ticagrelor
  Arms: Copayment Intervention Arm

SUMMARY:
Current patterns of P2Y12 receptor inhibitor use provide an excellent opportunity to test the impact of copayment reduction on clinician choice of medication, patient adherence, and clinical outcomes. The ARTEMIS trial is a practical multicenter, cluster- randomized clinical trial that will assess the impact of copayment reduction by equalizing the copayment of clopidogrel and ticagrelor. ARTEMIS will assess prescribing patterns, patient medication adherence, and clinical outcomes up to one year. We hypothesize that reducing out--of--pocket cost for P2Y12 receptor inhibitor will lead to improved adherence. Additionally, copayment reduction of both generic and brand antiplatelet agents may lead to a reduction in MACE risk. This is in part due to greater adherence to an evidence--based secondary prevention medication. Additionally the reduction in MACE may reflect greater selection of a more potent antiplatelet agent that has been shown to reduce MACE in randomized clinical trials, as provider choice of antiplatelet therapy will be primarily driven by risk- benefit assessment rather than the cost burden to the patient.

DETAILED DESCRIPTION:
ARTEMIS is a prospective, cluster-randomized clinical trial that will evaluate whether patient copayment elimination significantly influences antiplatelet therapy selection and long-term adherence, as well as patient outcomes and overall cost of care after acute myocardial infarction. Approximately 11,000 patients with ST-elevation myocardial infarction (STEMI) or non-STEMI (NSTEMI) will be enrolled at the approximately 300 hospitals in this study. Study sites selected for ARTEMIS will be geographically diverse, and will represent a diversity of hospital types and capabilities (e.g., teaching hospital, community hospital, etc). After institutional review board (IRB) approval of the study, each hospital will be randomized into either the intervention arm or the control arm. Hospitals randomized to the intervention arm will have the opportunity to offer enrolled patients either clopidogrel (generic P2Y12 receptor inhibitor option) or ticagrelor (brand P2Y12 receptor inhibitor option) without patient contribution to copayment in the next 12 months after the index MI discharge. Hospitals in the control arm will provide care per usual clinical routine. Notably, for both intervention and control arms, all patient management decisions (including the choice of antiplatelet therapy) are completely at the discretion of the care providers. Duration of antiplatelet therapy will also be at the discretion of care providers. All enrolled patients will be followed up to 15 months after index MI discharge to collect data on longitudinal treatment patterns and outcomes. Primary and secondary endpoints will be assessed at 12 months. An additional three months of follow up will assess for antiplatelet persistence and clinical events after discontinuation of the copayment intervention. Centralized follow-up will be conducted every 3 months via telephone or web-based contact.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study if they meet all of the following criteria:

* are ≥ 18 years of age
* have been diagnosed with STEMI or NSTEMI during the index hospitalization
* be treated with a P2Y12 receptor inhibitor at the time of enrollment
* have U.S. based health insurance coverage with prescription drug benefit
* have been fully informed and are able to provide written consent for longitudinal follow-up

Exclusion Criteria:

Patients are excluded if they meet any of the following criteria:

* have a history of prior intracranial hemorrhage
* have any contraindications to P2Y12 receptor inhibitor therapy at discharge
* involvement in another research study that specifies the type and duration of P2Y12 receptor inhibitor use within the next 12 months.
* have a life expectancy of less than one year
* have plans to move outside the US in the next year

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11001 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Wang, MD, MHS, MSc, Principal Investigator — Duke University; Eric Peterson, MD, MPH, FAHA, FACC, Study Chair — Duke University
Locations (228):
- United States (227):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Cottonwood, Arizona
  - Research Site, Flagstaff, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Fayetteville, Arkansas
  - Research Site, Fort Smith, Arkansas
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Escondido, California
  - Research Site, Huntington Beach, California
  - Research Site, Loma Linda, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Pasadena, California
  - Research Site, Riverside, California
  - Research Site, Salinas, California
  - Research Site, Stockton, California
  - Research Site, Thousand Oaks, California
  - Research Site, Torrance, California
  - Research Site, Vista, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Danbury, Connecticut
  - Research Site, New Haven, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Hudson, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Jacksonville Beach, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Largo, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orlando, Florida
  - Research Site, Panama City, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Cumming, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Suwanee, Georgia
  - Research Site, Honolulu, Hawaii
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Aurora, Illinois
  - Research Site, Belleville, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Joliet, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Urbana, Illinois
  - Research Site, Bloomington, Indiana
  - Research Site, Englewood, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Richmond, Indiana
  - Research Site, South Bend, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Davenport, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Overland Park, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Bossier City, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Rockport, Maine
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Clinton, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Salisbury, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Brighton, Massachusetts
  - Research Site, Hyannis, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Alpena, Michigan
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bay City, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Grand Blanc, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Jackson, Michigan
  - Research Site, Marquette, Michigan
  - Research Site, Mount Clemens, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Saint Joseph, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Warren, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Hattiesburg, Mississippi
  - Research Site, Bridgeton, Missouri
  - Research Site, Fenton, Missouri
  - Research Site, Joplin, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, North Kansas City, Missouri
  - Research Site, Saint Charles, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Billings, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, Flemington, New Jersey
  - Research Site, Haddon Heights, New Jersey
  - Research Site, Moorestown, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Paterson, New Jersey
  - Research Site, Pomona, New Jersey
  - Research Site, Ridgewood, New Jersey
  - Research Site, Teaneck, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albany, New York
  - Research Site, Cooperstown, New York
  - Research Site, Johnson City, New York
  - Research Site, New York, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Rochester, New York
  - Research Site, Schenectady, New York
  - Research Site, Staten Island, New York
  - Research Site, Stony Brook, New York
  - Research Site, Utica, New York
  - Research Site, Valhalla, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, High Point, North Carolina
  - Research Site, Lumberton, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Grand Forks, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Tualatin, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Allentown, Pennsylvania
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Chambersburg, Pennsylvania
  - Research Site, Danville, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Scranton, Pennsylvania
  - Research Site, Sellersville, Pennsylvania
  - Research Site, West Reading, Pennsylvania
  - Research Site, Wilkes-Barre, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Warwick, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Greenwood, South Carolina
  - Research Site, West Columbia, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, New Braunfels, Texas
  - Research Site, Palestine, Texas
  - Research Site, Plano, Texas
  - Research Site, Round Rock, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Temple, Texas
  - Research Site, Waco, Texas
  - Research Site, Webster, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Charlottesville, Virginia
  - Research Site, Lynchburg, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Roanoke, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Puyallup, Washington
  - Research Site, Renton, Washington
  - Research Site, Spokane, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Green Bay, Wisconsin
  - Research Site, La Crosse, Wisconsin
  - Research Site, Milwaukee, Wisconsin
  - Research Site, Racine, Wisconsin
  - Research Site, Waukesha, Wisconsin
- Research Site, Caguas, Puerto Rico

REFERENCES:
- [Derived] Rymer JA, Wegermann ZK, Kaltenbach LA, Webb LE, Peterson ED, Wang TY. Challenge in Predicting Persistence to P2Y12 Inhibitors: A Perspective From the ARTEMIS Trial. J Am Heart Assoc. 2023 Jun 20;12(12):e029063. doi: 10.1161/JAHA.122.029063. Epub 2023 Jun 10. PMID 37301758
- [Derived] Rymer JA, Kaltenbach LA, Peterson ED, Cohen DJ, Fonarow GC, Choudhry NK, Henry TD, Cannon CP, Wang TY. Does the Effectiveness of a Medicine Copay Voucher Vary by Baseline Medication Out-Of-Pocket Expenses? Insights From ARTEMIS. J Am Heart Assoc. 2022 Oct 18;11(20):e026421. doi: 10.1161/JAHA.122.026421. Epub 2022 Oct 17. PMID 36250667
- [Derived] Fanaroff AC, Peterson ED, Kaltenbach LA, Anstrom KJ, Fonarow GC, Henry TD, Cannon CP, Choudhry NK, Cohen DJ, Atreja N, Bhalla N, Eudicone JM, Wang TY. Copayment Reduction Voucher Utilization and Associations With Medication Persistence and Clinical Outcomes: Findings From the ARTEMIS Trial. Circ Cardiovasc Qual Outcomes. 2020 May;13(5):e006182. doi: 10.1161/CIRCOUTCOMES.119.006182. Epub 2020 May 12. PMID 32393129
- [Derived] Doll JA, Kaltenbach LA, Anstrom KJ, Cannon CP, Henry TD, Fonarow GC, Choudhry NK, Fonseca E, Bhalla N, Eudicone JM, Peterson ED, Wang TY. Impact of a Copayment Reduction Intervention on Medication Persistence and Cardiovascular Events in Hospitals With and Without Prior Medication Financial Assistance Programs. J Am Heart Assoc. 2020 Apr 21;9(8):e014975. doi: 10.1161/JAHA.119.014975. Epub 2020 Apr 17. PMID 32299284
- [Derived] Fanaroff AC, Peterson ED, Kaltenbach LA, Cannon CP, Choudhry NK, Henry TD, Anstrom KJ, Cohen DJ, Fonseca E, Khan ND, Fonarow GC, Wang TY. Agreement and Accuracy of Medication Persistence Identified by Patient Self-report vs Pharmacy Fill: A Secondary Analysis of the Cluster Randomized ARTEMIS Trial. JAMA Cardiol. 2020 May 1;5(5):532-539. doi: 10.1001/jamacardio.2020.0125. PMID 32129795
- [Derived] Fanaroff AC, Peterson ED, Kaltenbach LA, Cannon CP, Choudhry NK, Henry TD, Anstrom KJ, Cohen DJ, Fonseca E, Khan ND, Fonarow GC, Wang TY. Association of a P2Y12 Inhibitor Copayment Reduction Intervention With Persistence and Adherence With Other Secondary Prevention Medications: A Post Hoc Analysis of the ARTEMIS Cluster-Randomized Clinical Trial. JAMA Cardiol. 2020 Jan 1;5(1):38-46. doi: 10.1001/jamacardio.2019.4408. PMID 31721978
- [Derived] Wang TY, Kaltenbach LA, Cannon CP, Fonarow GC, Choudhry NK, Henry TD, Cohen DJ, Bhandary D, Khan ND, Anstrom KJ, Peterson ED. Effect of Medication Co-payment Vouchers on P2Y12 Inhibitor Use and Major Adverse Cardiovascular Events Among Patients With Myocardial Infarction: The ARTEMIS Randomized Clinical Trial. JAMA. 2019 Jan 1;321(1):44-55. doi: 10.1001/jama.2018.19791. PMID 30620370
- See also: D5130R00030_CSP_redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3805&filename=ARTEMIS%20D5130R00030_Protocol_03.12.2015%20REDACTED%20PDF.A.pdf
- See also: D5130R00030_SAP_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3805&filename=ARTEMIS_D5130R00030_SAP_Final_2017.11.30_signed_Redacted.PDF.A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruited patients on P2Y12 inhibitor therapy with US-based health insurance. Recruitment into 301 study sites (hospitals) in the US was conducted from June, 2015 to September, 2016. The study evaluated whether patient copayment reduction significantly influenced antiplatelet therapy selection and long-term adherence.
Pre-assignment Details: The study population included patients STEMI or NSTEMI who were treated with a P2Y12 receptor inhibitor. After patient enrollment into hospitals, each hospital was randomized into either the intervention or the control arm (cluster randomization). The randomization scheme was changed from 1:1 to 2:1 mid-study. 12 month study duration.
Period: Overall Study
Arm/Group | Copayment Intervention Arm | Usual Care Arm
Started (Total Patients Enrolled) | 6436 | 4565
Completed | 6135 | 3967
Not Completed | 301 | 598
Not completed — Death | 16 | 8
Not completed — Discharged without P2Y12 | 1 | 3
Not completed — Discharged on prasugrel | 283 | 587
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population for the primary analysis consists of all enrolled patients who survived the index MI hospitalization and did not withdraw before being discharged on clopidogrel or ticagrelor.
Groups:
- Total: Total of all reporting groups
Arm/Group | Copayment Intervention Arm | Usual Care Arm | Total
Number analyzed (Participants) | 6135 | 3967 | 10102
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Primary Population
  Years
    Age | 62.08 (11.78) | 62.10 (11.55) | 62.09 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender Population: Primary Population
  Participants
    Female | 1942 | 1285 | 3227
    Male | 4193 | 2682 | 6875
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity (Hispanic or Latino) Population: Primary Population
  Participants
    Hispanic or Latino | 188 | 222 | 410
    Not Hispanic or Latino | 5947 | 3745 | 9692
    Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race (White vs. Non-White)
  Participants
    Race: White | 5495 | 3416 | 8911
    Race: Non-White | 640 | 551 | 1191
Insurance Payors - Private Health Insurance [Count of Participants; unit: Participants] — Patients who have private health insurance Population: Primary Population
  Participants | 3864 | 2540 | 6404

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Cumulative Incidence Rate of Major Adverse Cardiovascular Events
Description: To determine if patient copayment reduction leads to lower risk of MACE (composite of death, MI, and stroke) at 1 year after discharge.
Time Frame: 12 months
Population: Primary Population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Copayment Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 6135 | 3967
Percentage of Participants | 10.17 [9.4 to 10.93] | 10.93 [9.67 to 11.60]
Statistical Analysis 1: Comparison: Copayment Intervention Arm vs Usual Care Arm; Test type: Superiority; p = 0.3503, Regression, Cox; Cox proportional hazards model accounting for within hospital clustering using robust standard errors; Hazard Ratio (HR) = 1.073, 95% CI 2-sided [0.925 to 1.246] — Usual Care arm is the reference group

2. Primary Outcome: Percentage of Patients With Long Term Non-persistence to P2Y12 Receptor Inhibitor
Description: To determine if patient copayment reduction leads to higher long-term persistence of any P2Y12 receptor inhibitor at 1 year after discharge.
Time Frame: 12 months
Population: Primary Population
Measure: Number; unit: Percentage of Patients
Arm/Group | Copayment Intervention Arm | Usual Care Arm
Number analyzed (Participants) | 6135 | 3967
Percentage of Patients | 12.96 | 16.21
Statistical Analysis 1: Comparison: Copayment Intervention Arm vs Usual Care Arm; Test type: Superiority; p = 0.0260, Regression, Logistic; Logistic regression model with parameters estimated using GEE to account for within hospital clustering for selected patient characteristics; Odds Ratio (OR) = 0.838, 95% CI 2-sided [0.717 to 0.979]

3. Secondary Outcome: P2Y12 Receptor Inhibitor Selection
Description: To evaluate whether reducing patient copayments for both generic and brand P2Y12 receptor inhibitor options affects medication selection at discharge.
Time Frame: 12 months
Population: Primary Population
Measure: Number; unit: Percentage of Patients
Groups:
- Copayment Intervention Arm - Clopidogrel: Patients in the intervention arm discharged on Clopidogrel
- Copayment Intervention Arm - Ticagrelor: Patients in the intervention arm discharged on Ticagrelor
- Usual Care Arm - Clopidogrel: Patients in the Usual Care Arm discharged on Clopidogrel
- Usual Care Arm - Ticagrelor: Patients in the Usual Care Arm discharged on Ticagrelor
Arm/Group | Copayment Intervention Arm - Clopidogrel | Copayment Intervention Arm - Ticagrelor | Usual Care Arm - Clopidogrel | Usual Care Arm - Ticagrelor
Number analyzed (Participants) | 6135 | 6135 | 3967 | 3967
Percentage of Patients | 36.0 | 59.6 | 54.7 | 32.4
Statistical Analysis 1: Comparison: Copayment Intervention Arm - Clopidogrel vs Copayment Intervention Arm - Ticagrelor vs Usual Care Arm - Clopidogrel vs Usual Care Arm - Ticagrelor; Test type: Superiority; p < 0.0001, Regression, Logistic; Logistic regression with GEE to account for within hospital clustering; Odds Ratio (OR) = 2.035, 95% CI 2-sided [1.564 to 2.649]

ADVERSE EVENTS:
Time Frame: Safety data was not actively collected in the ARTEMIS trial for the following reasons: • The safety profile of Brilinta (ticagrelor) is well established • ARTEMIS is a non-indication seeking interventional study that did not include a safety objective; the intervention involved co-payment only. Only Deaths were collected over the course of the 15-month study period.
Description: Adverse Events were only assessed with respect to All-Cause Mortality.
Arm/Group | Copayment Intervention Arm | Usual Care Arm
All-Cause Mortality (participants affected / at risk) | 16/6135 | 8/3967
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
1. Imbalances in enrollment and patient characteristics were expected in this cluster-randomized design due to differential incentives to enroll.
2. The cluster-randomized design renders the usual care arm vulnerable to potential bias to the null.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Registry Site shall submit to the Committee for its review a copy of any proposed publication resulting from the Registry at least thirty (30) days prior to the date of submission for publication or at least fifteen (15) days prior to submission for an abstract, and if no response is received within sixty (60) days of the date submitted to Sponsor, it will be conclusively presumed that the publication may proceed without delay.

DOCUMENTS (2):
  • Study Protocol (2015-03-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT02406677/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT02406677/SAP_001.pdf